CLINICAL TRIAL: NCT06821828
Title: Assessing Modified Olfactory Training to Prevent Cognitive Decline in MCI High-Risk Individuals: A Randomized Controlled Trial Protocol
Brief Title: The Efficacy of Modified Olfactory Training for MCI High-Risk Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Dawei Wu, Associate Researcher, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 9059101
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Subjective Cognitive Decline (SCD); Olfactory Dysfunction; Mild Cognitive Impairment (MCI); ELDERLY PEOPLE
Keywords: Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD); olfactory training; elderly population; Olfactory Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the Modified Olfactory Training Group (Experimental): Participants will use a modified olfactory training device based on expiratory pressure. Four odors will be used: rose, mint, lemon, and clove. Each odorant is sniffed for 10 seconds per session, with a 10-second interval between odors. Each training session lasts 5 minutes and is conducted twice daily, before breakfast and at bedtime, for a duration of two years.
  Interventions: Combination Product: Modified olfactory training device
- the Conventional Training Group (Active Comparator): Patients will receive the conventional olfactory training device. Patients had to sniff one odor for approximately 10 seconds and turn to another after a rest of 10 seconds. Each training session lasts 5 minutes and is conducted twice daily, before breakfast and at bedtime, for a duration of two years.
  Interventions: Combination Product: Conventional olfactory training device
- the Control Group (No Intervention): Participants will not receive any olfactory training and will be advised to observe and wait for spontaneous recovery of olfactory function.

INTERVENTIONS:
Combination Product: Modified olfactory training device — Participants will use a modified olfactory training device based on expiratory pressure. The advantages of the improved device are as follows: bi-directional airflow, positive pressure and the function of voice prompts and automatic counting.
  Arms: the Modified Olfactory Training Group
Combination Product: Conventional olfactory training device — This device involves four brown glass jars (total volume 5 mL) with one of the four odors in each (1mL each, soaked in cotton pads to prevent spilling). The following odors were used: phenyl ethyl alcohol (PEA): rose, menthol: mint, citronellal: lemon, and eugenol: cloves. All jars were labeled with the odor name.
  Arms: the Conventional Training Group

SUMMARY:
The goal of this clinical trial is to validate the effectiveness of the modified olfactory training device, the main questions it aims to answer are: Is it possible that the device can delay the progression of MCI in older adults? Compared to the conventional device, how efficient is the modified olfactory training device for improving cognitive function?

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) represents an intermediary stage between normal aging and dementia, with a significant proportion of cases progressing to dementia. No simple and effective therapeutic strategies are available to halt or reverse this progression. Olfactory dysfunction, a common early clinical manifestation of neurodegenerative diseases such as Alzheimer's Disease (AD), often precedes cognitive decline. Subjective Cognitive Decline (SCD) is increasingly recognized as a prodromal stage of MCI and dementia, which, together with olfactory dysfunction, provides a critical window for early intervention.

Conventional olfactory training (COT) has been shown to improve olfactory function, cognitive abilities, and brain connectivity in healthy elderly individuals, suggesting its potential to enhance neuroplasticity. Preliminary studies indicate that modified olfactory training (MOT) may yield superior outcomes compared to COT, with higher rates of olfactory recovery and improved deposition in the olfactory fissure. However, the efficacy of MOT in delaying or preventing the progression of olfactory dysfunction to MCI remains unclear.

In this study, the investigators planned to recruit 114 patients and divided them into three groups for control group and olfactory training with conventional and modified devices, and validate the effectiveness of the modified device based on changes in cognitive function and the comparison of the outcomes of the three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Gender: Individuals aged 60-80 years, regardless of gender.
2. Diagnosis of Idiopathic Olfactory Dysfunction: overall TDI score below 30.75 points using the Sniffin' Sticks test. Without olfactory impairment due to traumatic, sinusitis-related, congenital, toxic/drug-induced causes, post-operative conditions, tumors, or post-upper respiratory infections.
3. Diagnosis of Subjective Cognitive Decline: Montreal Cognitive Assessment (MoCA) score >24 for middle school level and above, >19 for elementary school level, and >13 for illiterate individuals. Amyloid β (Aβ) deposition in the brain (defined as Aβ42 < 550 ∼ 813 pg/ml)， the higher Formula of Hulstaert (defined as [(Aβ42/(240 + 1.18 × tau) ≤1]）, and hippocampus atrophy.
4. Consent: Willingness to sign an informed consent form.

Exclusion Criteria:

1. Comorbid Chronic Diseases or Severe Concurrent Illnesses: Individuals with conditions such as hypertension, diabetes, bronchopneumonia, malignant tumors， or chronic obstructive pulmonary disease.

4. Recent Medication Use: Exclusion of participants who have taken corticosteroids, antimicrobials, leukotriene antagonists, or antihistamines within the last four weeks.

5. Inability to Comply with Study Requirements: Based on the researcher's judgment, individuals who are unable to tolerate olfactory function tests and treatment， complete the study or comply with its requirements due to memory or behavioral abnormalities, depression, severe alcohol consumption, or previous non-compliance.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-03-22 (Estimated); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-05-22 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) score | Baseline,Month 3,Month 6,Month 12,Month 24
  The MoCA score will be used to evaluate cognitive function across several domains including memory, attention, language, and orientation.
Biomarkers of cognition (Blood/CSF) | Baseline,Month 3,Month 6,Month 12,Month 24
  This measure includes plasma and CSF levels of UGOT p-tau217, CSF Aβ42, p-tau181, total tau, and amyloid β 42 to total tau ratios. These biomarkers will help in assessing the biochemical progression of cognitive impairment.
Neuroimaging assessments | Baseline,Month 3,Month 6,Month 12,Month 24
  This includes MRI scans focusing on temporal lobes and other brain regions, and amyloid PET scans to detect amyloid plaques. These imaging techniques will provide insights into structural and functional changes in the brain associated with cognitive decline.
The Sniffin' Sticks test | Baseline,Month 3,Month 6,Month 12,Month 24
  a clinically significant olfactory improvement as measured by Sniffin' Sticks threshold, discrimination, and identification（TDI)( more than 6 scores)

SECONDARY OUTCOMES:
Auditory Verbal Learning Test (AVLT) | Baseline,Month 3,Month 6,Month 12,Month 24
  Evaluates immediate memory recall, learning rate, and delayed recall, providing insights into verbal learning and memory.
Digit Span Test (DST) | Baseline,Month 3,Month 6,Month 12,Month 24
  Assesses attention and working memory through forward and backward number recall tasks.
Trail Making Test (TMT) | Baseline,Month 3,Month 6,Month 12,Month 24
  Measures visual attention and task switching by requiring participants to connect a sequence of numbers and letters as quickly as possible.
Clock Drawing Test (CDT) | Baseline,Month 3,Month 6,Month 12,Month 24
  Used to assess visual-spatial abilities and executive function by having participants draw a clock showing a specific time.
Boston Naming Test (BNT) | Baseline,Month 3,Month 6,Month 12,Month 24
  Measures language function, specifically object naming ability, which is crucial for everyday communication.
Verbal Fluency Test (VFT) | Baseline,Month 3,Month 6,Month 12,Month 24
  Assesses cognitive flexibility and semantic memory by requiring participants to generate as many words as possible from a category in a limited time.
Activities of Daily Living Scale (ADL) | Baseline,Month 3,Month 6,Month 12,Month 24
  Evaluates the participant's ability to perform everyday tasks independently, reflecting functional status.
Instrumental Activities of Daily Living (IADL) | Baseline,Month 3,Month 6,Month 12,Month 24
  Assesses more complex daily living skills critical for independent living, such as managing finances and medication.
Neuropsychiatric Inventory (NPI) | Baseline,Month 3,Month 6,Month 12,Month 24
  Measures behavioral changes including depression, anxiety, aggression, and apathy among others, providing a comprehensive overview of psychological status.
Hamilton Anxiety Scale (HAMA) | Baseline,Month 3,Month 6,Month 12,Month 24
  Assesses the severity of anxiety symptoms, which can impact cognitive and daily functioning.
Hamilton Depression Scale (HAMD) | Baseline,Month 3,Month 6,Month 12,Month 24
  Used to quantify the level of depressive symptoms, aiding in the assessment of mood disorders which can co-occur with cognitive decline.
Olfactory bulb volume | Baseline,Month 3,Month 6,Month 12,Month 24
  Measurement of the olfactory bulb volume using MRI to assess changes or improvements in olfactory structures which might correlate with training efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Dawei Wu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will decide whether to share the individual participant data after the study.

REFERENCES:
- [Derived] Lin CY, Tan Y, Zhao D, Wu D. Assessing modified olfactory training to prevent cognitive decline in MCI high-risk individuals: a multicentre randomised controlled trial protocol in Beijing tertiary hospitals. BMJ Open. 2025 Aug 13;15(8):e100880. doi: 10.1136/bmjopen-2025-100880. PMID 40812823